CLINICAL TRIAL: NCT03047980
Title: Trial of Sirolimus for Cognitive Impairment in Sturge-Weber Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anne Comi, MD (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); Pfizer (Industry); National Institutes of Health (NIH) (NIH); Faneca 66 Foundation (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Anne Comi, MD, Principal Investigator, Director Sturge-Weber Center, Kennedy Krieger Institute, Professor Johns Hopkins University School of Medicine, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Organization: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00079722; 2U54NS065705 (NIH); BVMC6209 (Other Grant/Funding Number: Rare Diseases Clinical Research Network)
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Sturge-Weber Syndrome
Keywords: SWS; Cognitive impairment; sirolimus
MeSH Terms: conditions — Sturge-Weber Syndrome; Cognitive Dysfunction | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sirolimus (Experimental): All subjects will receive the sirolimus oral solution to be taken at home twice daily and will be treated on an outpatient basis. The drug will be taken for six months.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Low dose oral sirolimus
  Other Names: Rapamycin; Rapamune

SUMMARY:
The purpose of this research study is to gain a preliminary understanding of the safety of sirolimus in Sturge-Weber syndrome (SWS) and determine best outcomes to be used to assess the utility of sirolimus for the treatment of cognitive impairments related to Sturge-Weber syndrome.

DETAILED DESCRIPTION:
Sirolimus will be administered as an adjunct to all current medications. The impact of sirolimus upon cognitive functioning in Sturge-Weber syndrome is the primary outcome measure. This outcome will be assessed using a panel of testing selected based upon extensive experience in testing cognitive function in adults and children with SWS at the Kennedy Krieger Sturge-Weber Center. Changes in a quantitative EEG before and after the trial, Sturge-Weber syndrome clinical neuroscore, port-wine birthmark score, and the impact of sirolimus upon seizures will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages 3 to 31 years of age, inclusive.
2. Cognitive impairment as defined by the following:

   SWS cognitive neuroscore of ≥ 1
3. Ability to participate in direct neuropsychological and developmental testing.
4. English as primary language.
5. Stable anti-epileptic drugs (no changes in medications except dose for >3 months).
6. Adequate renal function. GFR must be greater than 50 ml/min/m2 as determined by the Schwartz Formula for children and MDRD for adults: http://www.nkdep.nih.gov/professionals/gfr_calculators/index.htm
7. If female and of child bearing potential, documentation of a negative pregnancy test prior to enrollment determined by a urine test is required. Sexually active pre-menopausal female patients (and female partners of male patients) must use adequate contraceptive measures, excluding estrogen containing contraceptives, while on the study drug. Abstinence will be considered an adequate contraceptive measure.
8. INR ≤1.5 (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks.)
9. Adequate liver function as shown by:

   * Serum bilirubin ≤ 1.5x ULN
   * ALT and AST ≤ 2.5x ULN
10. Written informed consent according to local guidelines. Local guidelines for subject assent will also be followed.
11. Stable dose of medications affecting the cytochrome P 450 3A4 (CYP3A4) and p glycoprotein (P gp) systems for at least 3 months prior to consent.

Exclusion Criteria:

1. Allergy to sirolimus or other rapamycin analogues.
2. Patients with seizures secondary to metabolic, toxic, infectious or psychogenic disorder, drug abuse or current seizures related to an acute medical illness.
3. Inability to keep follow-up appointments, maintain close contact with Principal Investigators, and/or complete all necessary studies to maintain safety.
4. Patients in need of immediate major surgical intervention.
5. Concurrent severe and/or uncontrolled medical disease, which could compromise participation in the pilot study (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration, impaired or restrictive pulmonary function, pneumonitis or pulmonary infiltrates).
6. Chronic treatment with systemic steroids or another immunosuppressive agent. Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary. Inhaled steroids are allowed.
7. Known history of HIV seropositivity or known immunodeficiency. Testing is not required unless a condition is suspected.
8. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of sirolimus (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection). A gastric tube or nasogastric tube is allowed.
9. Patients with an active, bleeding diathesis.
10. Patients with uncontrolled hyperlipidemia: fasting serum cholesterol > 300 mg/dL AND fasting triglycerides > 2.5 x ULN.
11. Patients who have had a major surgery or significant traumatic injury within four weeks of study entry. Patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the pilot study.
12. Patients with a prior history of organ transplant.
13. Patients who have received live attenuated vaccines within one week of start of sirolimus and during the pilot study.
14. Patients who have a history of malignancy.
15. Patients who are currently part of or have participated in any clinical investigation with an investigational drug within one month prior to enrollment.
16. Patients being treated with felbamate, unless treatment has been continuous for ≥ one year.
17. Patients currently receiving anticancer therapies or who have received anticancer therapies within four weeks of study entry (including chemotherapy, radiation therapy, antibody based therapy, etc.).

Ages: 3 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01; Primary Completion 2019-06-04 (Actual); Study Completion 2020-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Comi, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- See also: Hunter Nelson Sturge-Weber Center Website — http://www.kennedykrieger.org/patient-care/patient-care-centers/sturge-weber-center

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants will receive oral sirolimus.
Period: Overall Study
Arm/Group | Sirolimus
Started | 10
Completed | 9
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.58 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function as Assessed by the National Institute of Health (NIH) Toolbox Cognitive Battery
Description: Change over six months in cognitive functioning in Sturge-Weber syndrome is the primary outcome measure. This outcome will be assessed using the NIH Toolbox Cognitive Battery, a panel of testing which includes the following measures:
  * the Flanker Inhibitory Control and Attention Test (executive function and attention)
  * the Dimensional Change Card Sort Test (executive function)
  * Picture Sequence Memory Test (episodic memory)
  * Oral Reasoning Recognition Test and Picture Vocabulary Test (language skills)
  * Pattern Comparison Processing Speed Test (processing speed)
  * List Sorting Working Memory Test (working memory)
  * 9-hole Peg Test (dexterity)
  * Grip Strength Test (grip strength) and
  * Patient-Reported Outcomes Measurement Information System (PROMIS) (self-report emotional functioning).
  These scores are rescaled to T scores (mean = 50, standard deviation (SD) = 10), referenced against the US population. Higher scores indicate better outcome. T scores only were analyzed.
Time Frame: Baseline and at 6 months on the study drug
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Sirolimus
Number analyzed (Participants) | 9
T score
  National Institute of Health Toolbox Vocabulary Baseline | 44.2 (12.5)
  National Institute of Health Toolbox Vocabulary Follow-up | 42.3 (12.3)
  National Institute of Health Toolbox Attention Baseline | 34.1 (10.5)
  National Institute of Health Toolbox Attention Follow-up | 35.2 (14.1)
  National Institute of Health Toolbox Working Memory Baseline | 26.3 (9.8)
  National Institute of Health Toolbox Working Memory Follow-up | 28.1 (3.9)
  National Institute of Health Toolbox Executive Function Baseline | 33.1 (10.2)
  National Institute of Health Toolbox Executive Function Follow-up | 35.7 (15.4)
  National Institute of Health Processing Speed Baseline | 27.0 (14.5)
  National Institute of Health Processing Speed Follow-up | 36.4 (17.6)
  National Institute of Health Toolbox Sequential Memory Baseline | 39.3 (12.3)
  National Institute of Health Toolbox Sequential Memory Follow-up | 40.9 (8.6)
  National Institute of Health Toolbox Recognition Baseline | 37.7 (12.8)
  National Institute of Health Toolbox Recognition Follow-up | 36.0 (10.4)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Baseline | 43.5 (8.3)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Follow-up | 35.4 (20.5)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Baseline | 45.9 (7.9)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Follow-up | 35.7 (20.4)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Baseline | 53.8 (5.1)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Follow-up | 36.7 (15.3)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | 49.2 (11.1)
  Patient-Reported Outcomes Measurement Information System Pain (PROMIS) Interference Follow-up | 36.1 (18.8)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function Baseline | 46.9 (10.9)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Interference Follow-up | 41.9 (15.7)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Peer Relations Baseline | 49.8 (10.9)
  Patient-Reported Outcomes Measurement Information System (PROMIS) Peer Relations Follow-up | 44.1 (17.5)
  Grip Strength Dominant Baseline | 39.0 (14.4)
  Grip Strength Dominant Follow-up | 42.0 (5.1)
  Grip Strength Non-Dominant Baseline | 26.1 (28.2)
  Grip Strength Non-Dominant Follow-up | 20.6 (28.9)
  Dexterity Dominant Baseline | 30.6 (16.8)
  Dexterity Dominant Follow-up | 31.6 (14.3)
  Dexterity Non-Dominant Baseline | 31.6 (14.3)
  Dexterity Non-Dominant Follow-up | 30.1 (19.9)

2. Secondary Outcome: Difference in Mean Power Asymmetry of the Occipital Alpha Frequency Band
Description: Change in mean laterality score (by qEEG power analysis) was done comparing hemispheres and occipital lobes in the following frequency bands; delta, theta, alpha, beta, as previously described. As post-hoc analysis, baseline and follow-up qEEG of patients with and without stroke-like episodes were compared. Greater asymmetry with decreased power on the affected side is worse. We calculated a mean Laterality Score (LSb) for each band, averaged over 30 epochs and included channel pairs. Laterality Scores less than zero indicate lower power on the side ipsilateral to the port wine birthmark. In subjects who had a bilateral port wine birthmark, the side of maximal involvement was used (or the side of known involvement by MRI findings, where present).
Time Frame: Baseline and at 6months on the study drug
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus
Number analyzed (Participants) | 10
score on a scale
  Patients with Stroke-Like Episodes Baseline | 0.686 (0.03)
  Patients with Stroke-Like Episodes Follow-up | 0.426 (0.19)
  Patients without Stroke-like episodes Baseline | 0.167 (0.23)
  Patients without stroke-line episodes follow-up | 0.247 (0.13)

3. Secondary Outcome: Change in Sturge-Weber Syndrome Clinical Neuroscore
Description: Change in clinical neuroscore over the course of the study were measured. The neuroscore is comprised of frequency of seizures (0-4) , extent of hemiparesis (0-4), assessment of visual field cut (0-2) , and degree of cognitive functioning (0-5) with a minimum total score of 0 and a maximum total score of 15. Higher scores mean worsening of symptoms.
Time Frame: Baseline and at 6 months on the study drug
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Sirolimus
Number analyzed (Participants) | 10
score on a scale
  Composite Score Baseline | 4.5 [0 to 15]
  Composite Score Follow-up | 4.5 [0 to 15]
  Seizure Score Baseline | 1 [0 to 4]
  Seizure Score Follow-Up | 1 [0 to 4]
  Hemiparesis Score Baseline | 1 [0 to 4]
  Hemiparesis Score Follow-up | 1 [0 to 4]
  Visual Field Cut Score Baseline | 0.5 [0 to 2]
  Visual Field Cut Score Follow-up | 0 [0 to 2]
  Cognitive Function Score Baseline | 2.5 [0 to 5]
  Cognitive Function Score Follow-Up | 2.5 [0 to 5]

4. Secondary Outcome: Number of Participants With a Change in Sturge-Weber Syndrome Birthmark Score
Description: Frontal and profile photograph will be taken under standardized conditions with scoring of the port-wine birthmark for percent of face covered, thickness of birthmark, and darkness of birthmark color.
Time Frame: Visits at 2 weeks (baseline) and 28 weeks (study end)
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus
Number analyzed (Participants) | 10
Participants
  Improved Port-Wine Score | 4
  No Change Port-Wine Score | 2
  Worsened Port-Wine Score | 2
  No Port-Wine Birthmark | 2

ADVERSE EVENTS:
Time Frame: 6 months
Description: The Rare Diseases Clinical Research Network defines an adverse event as "...an unfavorable and unintended sign, symptom or disease associated with a participants' participation in a Rare Disease Clinical Research Network Study." The three types of adverse events are serious adverse events, unexpected adverse events and expected adverse events. This classification is using Common Terminology Criteria for Adverse Events developed and maintained by CTEP at National Cancer Institute.
Arm/Group | Sirolimus
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=10)
Headache (Nervous system disorders) | 1 (1) — Subject had a bad migraine with visual aura and was hospitalized on 9/27/2017. He was treated in the ER and hospitalized. Subject has a history of these events prior to going on study drug. This was deemed probably not related to the study drug.
Headache (Nervous system disorders) | 1 (1) — Subject developed a headache with vomiting and tingling/numbness on the left side. She experienced 2 brief focal seizures while in ER. This was probably not related to the study drug as the patient has a history of this event prior to study drug.
Anemia (Blood and lymphatic system disorders) | 1 (1) — Subject's final visit labs showed asymptomatic anemia with hemoglobin of 7.3. Patient had dark stools previously, making a GI bleed the likely source. She was off the study drug for 2 weeks prior so this is probably not related to the study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=10)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Skin Ulceration in Mouth (Skin and subcutaneous tissue disorders) | 3 (7)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Increased Alanine Aminotransferase (Investigations) | 1 (1)
Increased aspartate aminotransferase (Investigations) | 2 (3)
Cholesterol High (Investigations) | 1 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (9)
Decreased HDL Cholesterol (Investigations) | 2 (9)
Abnormal Urine Labs (Renal and urinary disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (4)
Seizure (Nervous system disorders) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
Personality Change (Product Issues) | 2 (2)
Behavioral Issues/ Aggression (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03047980/Prot_SAP_000.pdf